CLINICAL TRIAL: NCT07061834
Title: Enhancing Autonomic Regulation and Attention Through Galvanic Skin Response and Peripheral Temperature Biofeedback in Female Volleyball Players: a Randomized Pilot Trial
Brief Title: Enhancing Autonomic Regulation and Attention Through Biofeedback in Female Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Yucel Makaraci, Associate Professor, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMU_SBF-YM-01
Record Dates: First submitted 2025-07-01; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Psychological Aspects; Skin Temperature Change; Biofeedback Training; Volleyball Players; Autonomic Regulation
Keywords: Skin Conductance; biofeedback; mental health; attention; galvanic skin response
MeSH Terms: conditions — Psychological Well-Being | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: a parallel-group interventional design (biofeedback and control)
Masking Description: This study did not implement blinding or masking procedures for participants, investigators, or outcome assessors. Participants in both groups continued their regular volleyball training schedules; however, only the intervention group received the additional biofeedback training. The control group did not receive any specific treatment during the intervention period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback group (Experimental): The BFB group completed 15 sessions of multimodal BFB training over five weeks.
  Interventions: Device: Biofeedback training; Other: control group
- Control group (No Intervention): The control group received no intervention.

INTERVENTIONS:
Device: Biofeedback training — The intervention consists of biofeedback training using the Nexus 10 device, which provides real-time feedback on physiological signals including galvanic skin response and peripheral temperature. Participants undergo sessions where they learn to consciously regulate their autonomic nervous system activity by observing and modifying these signals. This training aims to improve stress regulation and enhance physiological self-control. Unlike other biofeedback interventions, this protocol focuses on combined skin conductance and temperature measures delivered through the Nexus 10 system over multiple sessions.
  Other Names: Multimodal biofeedback
  Arms: Biofeedback group
Other: control group — The control group received no intervention.
  Other Names: non intervention group
  Arms: Biofeedback group

SUMMARY:
This study aimed to evaluate the impact of a multimodal biofeedback intervention on autonomic function and sustained attention in female volleyball players.

DETAILED DESCRIPTION:
Optimal performance in elite athletes is shaped by a combination of physical preparedness and psychological readiness, where managing stress and anxiety is as critical as enhancing physical capabilities. Competitive anxiety can disrupt cognitive functioning, attention, and decision-making, affecting athletes' composure and overall performance. Cognitive abilities such as attentional control, mental flexibility, and perceptual-motor coordination are vital during high-pressure moments in sports, especially team sports like volleyball. Emerging approaches in applied sports psychology have started using biofeedback (BFB) to address these psychological and cognitive demands. BFB enables athletes to consciously regulate physiological responses associated with stress, such as heart rate variability (HRV), galvanic skin response (GSR), peripheral temperature (PT), and muscle activity, by providing real-time feedback. These interventions aim to enhance autonomic control, emotional regulation, and ultimately, cognitive performance.

Multimodal BFB interventions that simultaneously target several physiological parameters are gaining attention for their potential to support mental readiness and attentional performance in athletes. However, the application of such protocols in team sports remains underexplored. Given the high cognitive demands of volleyball, especially in sustained attention and rapid decision-making under pressure, there is a need to examine whether multimodal BFB can produce meaningful improvements in these areas. This study investigated the effects of a five-week, 15-session multimodal BFB intervention on sustained attention and physiological responses in competitive female volleyball players. It was hypothesized that the intervention would lead to measurable physiological changes-specifically a reduction in GSR and an increase in PT-which in turn would support improved cognitive performance in the form of enhanced sustained attention.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Nonsmoking status
* A history of regular menstrual cycles
* No mental, neurological, or cardiovascular disorders
* Active participation in national volleyball tournaments

Exclusion Criteria:

* Use of illegal substances, oral contraceptives, antidepressants
* Consuming alcohol or drugs
* Current psychotherapy
* A history of BFB intervention

Ages: 17 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Attention | From enrollment to the end of treatment at 5 weeks"
  Sustained Attention in this study was assessed using the d2 Test of Attention, a standardized paper-and-pencil test designed to measure an individual's ability to maintain focused and selective attention over a continuous period. During the test, participants were required to scan rows of letters and quickly identify and mark the target letter "d" with two dashes, while ignoring similar distracting stimuli. The test evaluates concentration, processing speed, and the ability to sustain attention under time pressure. Performance is quantified by the number of correctly identified targets minus errors, reflecting how effectively the participant can sustain attention and resist distractions throughout the task.

SECONDARY OUTCOMES:
Galvanic Skin Response | From enrollment to the end of treatment at 5 weeks.
  Galvanic Skin Response (GSR) refers to changes in the skin's electrical conductance, which vary with sweat gland activity and are linked to physiological arousal and emotional states. In this study, GSR was measured as a secondary outcome using biofeedback training with the Nexus 10 device, a system that records real-time skin conductance data through sensors placed on the participant's fingers. This measurement reflects the participant's autonomic nervous system activity, providing insight into stress levels, emotional regulation, and overall physiological responses during the biofeedback sessions.
Peripheral Temperature | From enrollment to the end of treatment at 5 weeks.
  Peripheral Temperature refers to the temperature of the skin on the extremities, such as fingers or toes, which can indicate changes in blood flow and autonomic nervous system activity. In this study, peripheral temperature was measured as a secondary outcome using the Nexus 10 device during biofeedback training. Sensors placed on the participant's fingers recorded skin temperature continuously, providing information about physiological responses related to relaxation, stress, and circulation.

CONTACTS AND LOCATIONS:
Overall Officials: Yücel Makaracı Makaracı, PhD, Study Director — Karamanoğlu Mehmetbey University
Locations (1):
- Faculty of Sports Sciences, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to protect participant privacy and because consent did not cover data sharing beyond the research team.

REFERENCES:
- [Derived] Makaraci M, Makaraci Y. Enhancing autonomic regulation and attention through galvanic skin response and peripheral temperature biofeedback in female volleyball players: a randomized pilot trial. BMC Sports Sci Med Rehabil. 2025 Sep 26;17(1):274. doi: 10.1186/s13102-025-01344-7. PMID 41013699
- See also: pubmed page — https://pubmed.ncbi.nlm.nih.gov/39149880/